CLINICAL TRIAL: NCT03846843
Title: An Open-Label, Two-Part, Phase 1/2a, Crossover Study to Determine the Absolute Bioavailability and Pharmacokinetics of Oral Immediate-Release Doses of OCR-002 in Subjects With Varying Degrees of Cirrhosis
Brief Title: OCR002-SP103 - Oral Immediate Release Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ocera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: OCR002-SP103
Record Dates: First submitted 2017-11-02; First posted 2019-02-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Cirrhosis
Keywords: Child-Pugh Class B
MeSH Terms: conditions — Fibrosis | interventions — ornithine phenylacetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- OCR-002 - Treatment A (Experimental): A single 5 g oral dose of OCR-002 oral solution administered under fasting conditions
  Interventions: Drug: OCR-002 Oral Solution
- OCR-002 - Treatment B (Experimental): A single 5 g oral dose of OCR-002 oral solution administered under fed conditions
  Interventions: Drug: OCR-002 Oral Solution
- OCR-002 - Treatment C (Experimental): A single 5 g intravenous dose of OCR-002 solution infused over 1 hour under fasting conditions
  Interventions: Drug: OCR-002 IV Solution
- OCR-002 - Treatment D (Experimental): A single 5 g oral dose of OCR-002 oral solution administered under fasting conditions following discontinuation of lactulose
  Interventions: Drug: OCR-002 IV Solution
- OCR-002 - Treatment E (Experimental): 6 g OCR-002 per day (2 tablets TID for 6 g total daily dose)
  Interventions: Drug: OCR-002 IR Oral Tablet
- OCR-002 - Treatment F (Experimental): 12 g OCR-002 per day (4 tablets TID for 12 g total daily dose)
  Interventions: Drug: OCR-002 IR Oral Tablet
- OCR-002 - Treatment G (Experimental): 21 g OCR-002 per day (7 tablets TID for 21 g total daily dose)
  Interventions: Drug: OCR-002 IR Oral Tablet

INTERVENTIONS:
Drug: OCR-002 IR Oral Tablet — OCR-002 3 gram immediate release (IR) tablet for oral administration
  Other Names: Ornithine phenylacetate
  Arms: OCR-002 - Treatment E; OCR-002 - Treatment F; OCR-002 - Treatment G
Drug: OCR-002 Oral Solution — OCR-002 5 gram solution for oral administration
  Other Names: Ornithine phenylacetate
  Arms: OCR-002 - Treatment A; OCR-002 - Treatment B
Drug: OCR-002 IV Solution — OCR-002 5 gram solution for intravenous (IV ) administration
  Other Names: Ornithine phenylacetate
  Arms: OCR-002 - Treatment C; OCR-002 - Treatment D

SUMMARY:
This is an open-label Phase 1, 2-part, crossover study in approximately 33 adult subjects (12 subjects in Part 1 and 21 subjects in Part 2), with varying degrees of cirrhosis with analysis of pharmacokinetic (PK) data after Part 1 to guide dose regimen selection and PK sampling time points for OCR-002 in Part 2.

DETAILED DESCRIPTION:
Part 1: Dosing Periods 1, 2, 3, and 4:

Single-dose, partially randomized, 4-period crossover study to evaluate 5 g OCR-002 oral solution administered under fed conditions, fasting conditions, or under fasting conditions following discontinuation of lactulose in 12 subjects with cirrhosis (Child-Pugh class A and C).

The purpose is to determine the pharmacokinetics of phenylacetic acid (PAA) and phenylacetylglutamine (PAGN) following a single 5 g dose of OCR-002 oral solution administered under fed conditions, fasting conditions, or under fasting conditions following discontinuation of lactulose as compared to a single 5 g intravenous dose of OCR-002 under fasting conditions in subjects with cirrhosis (Child-Pugh class A and C).

Analysis of pharmacokinetic data will be conducted after completion of Part 1 in order to determine the dose regimen of OCR-002 oral tablets to use in Part 2 of the study.

Part 2: Dosing Periods 1, 2 and 3:

Multiple-dose, randomized, 3-period crossover study to evaluate OCR-002 oral tablets in subjects with cirrhosis (Child-Pugh class B). The purpose is to characterize the PK and pharmacodynamic (PD) of OCR-002 tablets after TID administration for 5 days in subjects with cirrhosis (Child-Pugh class B).

ELIGIBILITY:
Inclusion Criteria

Subjects eligible for enrollment must meet all of the following inclusion criteria:

1. Informed of the nature of the study and provided written informed voluntary consent;
2. Male or female ≥18 years of age or the legal age of consent (whichever is greater) and ≤70 years of age at the time of Screening;
3. Willing and able to abstain from tobacco products and alcohol during confinement at the research unit;
4. Evidence of/known cirrhosis (Child-Pugh class A and C in Part 1, Child-Pugh class B in Part 2). Diagnosis of liver cirrhosis will be based on clinical, radiological, or histological criteria;
5. Currently using lactulose (minimum of 5 days prior to Day -1)
6. If using rifaximin at Screening Visit, it must be discontinued at least 7 days before the first dose of study drug;
7. Negative serum pregnancy test (females of childbearing potential only);
8. Agree to utilize an effective barrier method (mechanical barrier, intrauterine device, or condom with spermicide) of contraception from Screening through to at least 4 weeks after the last dose of study drug for sexually active female who is not surgically sterile or post-menopausal. Sexually active males must use contraception and also refrain from donating sperm while on study drug from admission to at least 4 weeks after the last dose of study drug; Able to communicate effectively with the Investigator/designee and other study center personnel and agree to comply with the study procedures and restrictions.

Exclusion Criteria

Subjects meeting any of the following criteria will not be eligible for enrollment:

1. Not expected to survive for 2 months;
2. Presence of Type 1 hepatorenal syndrome;
3. Presence of hyponatremia (serum sodium <125 mmol/L);
4. Presence of renal failure with serum creatinine >3 mg/dL or need for hemodialysis, peritoneal dialysis, or continuous venovenous hemofiltration at Screening;
5. New York Heart Association Class 3 or 4 congestive heart failure or overt clinical signs of congestive heart failure;
6. Requirement for mechanical ventilation (continuous positive airway pressure is allowed);
7. Prior transplant recipient (solid organ, bone marrow, or stem cell);
8. Any prior stroke with cognitive sequelae;
9. Presence of acute alcoholic hepatitis;
10. Positive test for human immunodeficiency virus or hepatitis B surface antigen;
11. Presence of overt hepatic encephalopathy, other irreversible brain damage, aspiration pneumonia, or severe psychiatric disorder;
12. Known or suspected gastrointestinal bleeding within 7 days before Screening;
13. Hemodynamic instability, defined as mean arterial blood pressure <60 mmHg and/or evidence of poor organ perfusion;
14. Current use of more than 1 vasopressor to support blood pressure;
15. Current use of drugs that could potentially interfere with renal excretion of PAGN, such as probenecid, estrone sulfate, ibuprofen, cimetidine, or diclofenac. Use of L-ornithine L-aspartate is prohibited;
16. Current use of drugs whose renal excretion may be affected by OCR-002, such as quinidine, metformin, or cimetidine;
17. Current use of molecular adsorbent recirculation system;
18. Current use of AMMONUL (sodium benzoate with sodium phenylacetate), BUPHENYL (sodium phenylbutyrate), RAVICTI, or other medications that contain sodium benzoate or sodium phenylbutyrate.
19. Current use of rifaximin or oral neomycin;
20. Corrected QT interval (Fridericia's formula) >480 msec at Day -1;
21. History or allergic reactions to ornithine, PAA, or their analogs;
22. Currently hospitalized for any reason or clinically significant surgery within 4 weeks before the first dose of the study drug;
23. Presence of transjugular intrahepatic portosystemic shunt;
24. Blood loss or blood donation of >500 mL within 30 days or plasma donation >500 mL within 14 days before administration of the first dose of study drug;
25. Currently lactating;
26. Positive screening result for drugs of abuse;
27. Ingestion of grapefruit or grapefruit juice within 48 hours before study dose administration; or use of repaglinide throughout the study;
28. Receipt of an investigational product or device, or participation in a drug research study within a period of 30 days (or 5 half-lives of the drug, whichever is longer) before the first dose of study drug;
29. Prior diagnosis of cancer and receiving active therapy, or hepatic cancer or cancer with known brain metastasis;
30. Any condition or set of circumstances which, in the judgment of the Investigator or Sponsor, could interfere with their ability to comply with the dosing schedule and completion of the study evaluations.
31. Prior surgical shunt recipient (Part 2)
32. Subject has a body weight <45 kg (Part 2).
33. Current use of oral vancomycin or oral or parenteral antibiotic that could potentially alter gut flora (Part 2)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of PAA and PAGN following described treatment | 6 months
  Maximum concentration (Cmax) of PAA and PAGN following a single 5 g dose of OCR-002 oral solution under fed or fasting conditions as compared to a single 5 g IV dose of OCR-002 under fasting conditions in participants with cirrhosis (Child-Pugh Classes A and C). Plasma concentrations of PAA, PAGN and ornithine will be analyzed by non-compartmental PK methods.
Time to Cmax (Tmax) of PAA and PAGN | 6 months
  Plasma concentrations of PAA, PAGN and ornithine will be analyzed by non-compartmental PK methods.
Area under the plasma concentration time curve over time (AUC0-t) of PAA and PAGN following described treatment | 6 months
  Area under the plasma concentration time curve over time (AUC0-t) of PAA and PAGN following a single 5 g dose of OCR-002 oral solution under fed or fasting conditions as compared to a single 5 g IV dose of OCR-002 under fasting conditions in participants with cirrhosis (Child-Pugh Classes A and C). Plasma concentrations of PAA, PAGN and ornithine will be analyzed by non-compartmental PK methods.
AUC0-24 of PAA and PAGN following a single 5 g dose of OCR-002 oral solution under fed or fasting conditions as compared to a single 5 g IV dose of OCR-002 under fasting conditions in participants with cirrhosis (Child-Pugh Classes A and C) | 6 months
  Plasma concentrations of PAA, PAGN and ornithine will be analyzed by non-compartmental PK methods.
AUC0-36 of PAA and PAGN following a single 5 g dose of OCR-002 oral solution under fed or fasting conditions as compared to a single 5 g IV dose of OCR-002 under fasting conditions in participants with cirrhosis (Child-Pugh Classes A and C) | 6 months
  Plasma concentrations of PAA, PAGN and ornithine will be analyzed by non-compartmental PK methods.
AUC0-inf of PAA and PAGN following a single 5 g dose of OCR-002 oral solution under fed or fasting conditions as compared to a single 5 g IV dose of OCR-002 under fasting conditions in participants with cirrhosis (Child-Pugh Classes A and C) | 6 months
  Plasma concentrations of PAA, PAGN and ornithine will be analyzed by non-compartmental PK methods.
Half-life (t1/2) of PAA and PAGN following a single 5 g dose of OCR-002 oral solution under fed or fasting conditions as compared to a single 5 g IV dose of OCR-002 under fasting conditions in participants with cirrhosis (Child-Pugh Classes A nd C) | 6 months
  Plasma concentrations of PAA, PAGN and ornithine will be analyzed by non-compartmental PK methods.
Evaluate the effect of a high-fat meal on the Cmax of 5 g OCR-002 oral solution in participants with cirrhosis (Child-Pugh Classes A and C) | 6 months
  Participants will fast overnight for at least 8 hours prior to receiving the high fat (approximately 50% of total calorie content of the meal) and high-calorie (approximately 800 to 1000 calories) test meal, which will be entirely consumed within 30 minutes or less.
Evaluate the effect of a high-fat meal on the AUC of 5 g OCR-002 oral solution in participants with cirrhosis (Child-Pugh Classes A and C) | 6 months
  Participants will fast overnight for at least 8 hours prior to receiving the high fat (approximately 50% of total calorie content of the meal) and high-calorie (approximately 800 to 1000 calories) test meal, which will be entirely consumed within 30 minutes or less.
Evaluate the effect of a high-fat meal on oral bioavailability of 5 g OCR-002 oral solution in participants with cirrhosis (Child-Pugh Classes A and C) | 6 months
  Participants will fast overnight for at least 8 hours prior to receiving the high fat (approximately 50% of total calorie content of the meal) and high-calorie (approximately 800 to 1000 calories) test meal, which will be entirely consumed within 30 minutes or less.
Cmax of PAA and PAGN following a single dose of OCR-002 oral solution under fasting conditions in participants with cirrhosis who have discontinued lactulose (Child-Pugh Classes A and C) | 6 months
  Cmax of PAA and PAGN following a single dose of OCR-002 oral solution under fasting conditions in participants with cirrhosis who have discontinued lactulose (Child-Pugh Classes A and C) will be determined.
AUC of PAA and PAGN following a single dose of OCR-002 oral solution under fasting conditions in participants with cirrhosis who have discontinued lactulose (Child-Pugh Classes A and C) | 6 months
  AUC of PAA and PAGN following a single dose of OCR-002 oral solution under fasting conditions in participants with cirrhosis who have discontinued lactulose (Child-Pugh Classes A and C) will be determined.
Urinary excretion of PAGN following a single dose of each treatment in participants with cirrhosis (Child-Pugh Classes A and C) | 6 months
  Urinary excretion profile of PAGN following a single dose of each treatment in participants with cirrhosis (Child-Pugh Classes A and C) will be determined.
Cmax of OCR-002 immediate-release tablets over the course of TID dosing for 5 days | 5 days
  Cmax of OCR-002 immediate-release tablets over the course of TID dosing for 5 days will be determined.
Cmax of PAA, PAGN, and ornithine following 3 times a day (TID) OCR 002 oral tablet administration for 5 days in participants with cirrhosis | 5 days
  Cmax of PAA, PAGN, and ornithine following 3 times a day (TID) OCR 002 oral tablet administration for 5 days in participants with cirrhosis will be determined.
Ammonia-lowering (Tmax) effect of OCR-002 over the course of TID dosing for 5 days | 5 days
  Ammonia-lowering (Tmax) effect of OCR-002 over the course of TID dosing for 5 days will be determined.
AUC of oral, immediate-release (IR) OCR 002 tablets | 5 days
  AUC of oral, immediate-release (IR) OCR 002 tablets will be determined.
AUC of PAA, PAGN, and ornithine following 3 times a day (TID) OCR 002 oral tablet administration for 5 days in participants with cirrhosis | 5 days
  AUC of PAA, PAGN, and ornithine following 3 times a day (TID) OCR 002 oral tablet will be determined.
Degree of fluctuation (Day 5) of OCR-002 immediate-release tablets | 5 days
  Degree of fluctuation (Day 5) of OCR-002 immediate-release tablets will be determined.
Elimination rate constant (kel) of OCR-002 immediate-release tablets | 5 days
  kel of OCR-002 immediate-release tablets will be determined.
T1/2 of OCR-002 immediate-release tablets | 5 days
  T1/2 of OCR-002 immediate-release tablets will be determined.
Drug elimination (Cmax) following discontinuation of OCR-002 oral tablets after TID administration for 5 days | 5 days
  Drug elimination (Cmax) following discontinuation of OCR-002 oral tablets will be determined.
Urinary excretion profile of urea following TID administration of OCR-002 oral tablets of each treatment in participants with cirrhosis | 5 days
  Urinary excretion profile of urea following TID administration of OCR-002 oral tablets of each treatment in participants with cirrhosis will be determined.
Urinary excretion of PAGN following TID administration of OCR 002 oral tablets of each treatment in participants with cirrhosis | 5 days
  Urinary excretion of PAGN following TID administration of OCR 002 oral tablets of each treatment in participants with cirrhosis will be determined
Urinary excretion of PAA following TID administration of OCR 002 oral tablets of each treatment in participants with cirrhosis | 5 days
  Urinary excretion of PAA following TID administration of OCR 002 oral tablets of each treatment in participants with cirrhosis will be determined.
Change from Baseline in serum blood urea nitrogen (BUN) over the course of TID dosing for 5 days | 5 days
  Change from Baseline in serum BUN over the course of TID dosing for 5 days will be calculated.
Change from Baseline in serum creatinine over the course of TID dosing for 5 days | 5 days
  Change from Baseline in serum creatinine over the course of TID dosing for 5 days will be calculated.
Change from Baseline in creatinine clearance over the course of TID dosing for 5 days | 5 days
  Change from Baseline in creatinine clearance over the course of TID dosing for 5 days will be calculated.
Urea clearance over the course of TID dosing for 5 days | 5 days
  Urea clearance over the course of TID dosing for 5 days will be calculated.
Percent of PAA dose excreted in urine as PAGN and unchanged (as PAA) over each collection interval and the entire collection interval | 5 days
  Percent of PAA dose excreted in urine as PAGN and unchanged (as PAA) over each collection interval and the entire collection interval will be calculated.

SECONDARY OUTCOMES:
Adverse events of 5 g OCR-002 oral solution in participants with cirrhosis (Child-Pugh class A and C) | 6 months
  Adverse events data will be summarized.
Adverse events of OCR-002 in participants with cirrhosis following multiple TID doses of OCR-002 tablets | 6 months
  Adverse events data will be summarized.
Change from Baseline in sitting blood pressure of 5 g OCR-002 oral solution in participants with cirrhosis (Child-Pugh class A and C) | 6 months
  Sitting blood pressure will be measured after the participant has been in a sitting position for at least 3 minutes.
Change from Baseline in heart rate of 5 g OCR-002 oral solution in participants with cirrhosis (Child-Pugh class A and C) | 6 months
  Heart rate will be measured after the participant has been in a sitting position for at least 3 minutes.
Change from Baseline in body temperature of 5 g OCR-002 oral solution in participants with cirrhosis (Child-Pugh class A and C) | 6 months
  Body temperature will be measured after the participant has been in a sitting position for at least 3 minutes.
Change from Baseline in sitting blood pressure of OCR-002 in participants with cirrhosis following multiple TID doses of OCR-002 tablets | 6 months
  Sitting blood pressure will be measured after the participant has been in a sitting position for at least 3 minutes.
Change from Baseline in heart rate of OCR-002 in participants with cirrhosis following multiple TID doses of OCR-002 tablets | 6 months
  Heart rate will be measured after the participant has been in a sitting position for at least 3 minutes.
Change from Baseline in body temperature of OCR-002 in participants with cirrhosis following multiple TID doses of OCR-002 tablets | 6 months
  Body temperature will be measured after the participant has been in a sitting position for at least 3 minutes.
Proportion of participants with abnormal clinical chemistry values of 5 g OCR-002 oral solution in participants with cirrhosis (Child-Pugh class A and C) | 6 months
  Treatment-emergent abnormal laboratory tests are those in which the baseline value is normal (within the laboratory normal reference range) and post-baseline value is abnormal (i.e., meets Grade III or Grade IV toxicity criteria from the National Cancer Institute Common Terminology Criteria.
Proportion of participants with abnormal hematology values of 5 g OCR-002 oral solution in participants with cirrhosis (Child-Pugh class A and C) | 6 months
  Treatment-emergent abnormal laboratory tests are those in which the baseline value is normal (within the laboratory normal reference range) and post-baseline value is abnormal (i.e., meets Grade III or Grade IV toxicity criteria from the National Cancer Institute Common Terminology Criteria.
Proportion of participants with abnormal clinical chemistry values of OCR-002 in participants with cirrhosis following multiple TID doses of OCR-002 tablets | 6 months
  Treatment-emergent abnormal laboratory tests are those in which the baseline value is normal (within the laboratory normal reference range) and post-baseline value is abnormal (i.e., meets Grade III or Grade IV toxicity criteria from the National Cancer Institute Common Terminology Criteria.
Proportion of participants with abnormal hematology values of OCR-002 in participants with cirrhosis following multiple TID doses of OCR-002 tablets | 6 months
  Treatment-emergent abnormal laboratory tests are those in which the baseline value is normal (within the laboratory normal reference range) and post-baseline value is abnormal (i.e., meets Grade III or Grade IV toxicity criteria from the National Cancer Institute Common Terminology Criteria.
Proportion of participants with abnormal urinalysis values of 5 g OCR-002 oral solution in participants with cirrhosis (Child-Pugh class A and C) | 6 months
  Treatment-emergent abnormal laboratory tests are those in which the baseline value is normal (within the laboratory normal reference range) and post-baseline value is abnormal (i.e., meets Grade III or Grade IV toxicity criteria from the National Cancer Institute Common Terminology Criteria.
Proportion of participants with abnormal urinalysis values of OCR-002 in participants with cirrhosis following multiple TID doses of OCR-002 tablets | 6 months
  Treatment-emergent abnormal laboratory tests are those in which the baseline value is normal (within the laboratory normal reference range) and post-baseline value is abnormal (i.e., meets Grade III or Grade IV toxicity criteria from the National Cancer Institute Common Terminology Criteria.
Cmax of ornithine over the course of TID administration of OCR-002 for 5 days | 5 days
  Cmax of ornithine over the course of TID administration of OCR-002 for 5 days will be reported.
Tmax of ornithine over the course of TID administration of OCR-002 for 5 days | 5 days
  Tmax of ornithine over the course of TID administration of OCR-002 for 5 days will be reported.
AUC0-24 of ornithine over the course of TID administration of OCR-002 for 5 days | 5 days
  AUC0-24 of ornithine over the course of TID administration of OCR-002 for 5 days will be reported.
Degree of fluctuation of ornithine over the course of TID administration of OCR-002 for 5 days | 5 days
  Degree of fluctuation of ornithine over the course of TID administration of OCR-002 for 5 days will be reported.
kel of ornithine over the course of TID administration of OCR-002 for 5 days | 5 days
  kel of ornithine over the course of TID administration of OCR-002 for 5 days will be reported.
T1/2 of ornithine over the course of TID administration of OCR-002 for 5 days | 5 days
  T1/2 of ornithine over the course of TID administration of OCR-002 for 5 days will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (1):
- Southern California Research Center, Coronado, California, United States

IPD SHARING:
Plan to Share IPD: No